CLINICAL TRIAL: NCT04083300
Title: 6-8 Years Follow up of Cancer Survivors, Objectively Measured Physical Activity and Quality of Life Over Time.
Brief Title: Cancer, Physical Activity and Quality of Life- a Longterm Follow up
Status: Completed | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2018/1788
Record Dates: First submitted 2019-06-18; First posted 2019-09-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2020-01

CONDITIONS: Cancer; Rehabilitation; Stress Disorder; Fatigue; Quality of Life; Physical Activity
MeSH Terms: conditions — Neoplasms; Stress Disorders, Traumatic; Fatigue; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project is a 6-8-years follow-up of a randomized controlled trial testing a stepped care stress management program. The main goal is to examining differences in long-term effects on cancer-related stress reactions and emotional reactivity between the intervention and control group. Secondary objectives is to investigate consequences of cancer and its' treatment over time, such as long term quality of life, objectively physical activity and experiences concerning follow-up and the transition from specialist health services to municipal health services.

DETAILED DESCRIPTION:
Major improvements in cancer detection and treatment lead to longer life expectancy among cancer survivors. This may in turn lead to more late effects and many have to deal with long-term consequences of the disease and its' treatment. Returning to everyday life and to work is often an important part of returning to normal life for cancer survivors. There is increasing knowledge concerning late effects, but there is still lack of knowledge concerning the life of those experiencing late effects. There is a need for more knowledge about late effects' impact on the return to work prosess, physical activity and quality of life over time. Both quantitative and qualitative methods will be utilized. Standardized questionnaires will provide information on the effect of the intervention over time, in addition to quality of life over time. Sensewear armband will provide information about their physical activity over time. Official register data from the Norwegian Labour and Welfare Administration (the NAV administration) will provide us information about the work- and benefit situation through the whole follow-up period of 6-8 years. The register data include information about type of social benefits (sick-leave benefit, work assessment allowance (WAA), disability pension, unemployment benefit and retirement pension), as well as information about occupation, income and sick leave diagnosis. Focus group interviews will give us insight in the cancer survivors own experiences with quality of life over time, the transition from the specialist health services to the primary health care and the follow-up in the municipalities.

ELIGIBILITY:
Inclusion Criteria:

* Stage I-III disease
* Scheduled for neo/adjuvant or curative treatment (i.e. chemotherapy, radiation therapy or hormonal therapy or any combination of these therapies)

Exclusion Criteria:

* On-going psychiatric condition
* Lack of fluency in Norwegian
* A previous diagnosis of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer survivors who participated in the early "Early rehabilitation of cancer patients" (ClinicalTrials.gov Identifier: NCT 01588262) were asked to join this follow up study.
Sampling Method: Probability Sample
Enrollment: 271 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Cancer-related stress reactions 6-8 years after the diagnosis and inclusion in the study. | 2021
Objectively measured physical activity from diagnosis to 6-8 years follow up. | 2022
The context between change in physical activity and quality of life over time | 2023
Witch predictors has an impact on long term cancer survivors quality of life? | 2024

SECONDARY OUTCOMES:
Cancer survivors' experience of quality of life 6-8 years after diagnosis- a qualitative study | 2021
  Experiences of the follow up.

OTHER OUTCOMES:
The participants ability to work during the 5-years follow-up, using official register data and questionnaires. | 2020
  How many patients have been receiving sickness benefits, full or partial, or have returned to work. What characterizes the participants that fell out of working life after the cancer disease, concerning factors such as quality of life and social inequality measured by The Hospital Anxiety and Depression Scale (A 14-item questionnaire, where >8 indicate clinically significant level of anxiety/depression).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology and Medical Physics, Cancer center for Education and rehabilitation, Haukeland University Hospital, Bergen, Norway